CLINICAL TRIAL: NCT06691763
Title: The Effect of Pythagorean Self-Awareness Technique on Patients with Psoriasis. the Alternations in Hair Cortisol Levels Via Affecting Hypothalamic-Pituitary-Adrenal Axis.
Brief Title: Pythagorean Self-Awareness Intervention on Psoriasis Patients.
Acronym: PSAIPSORIASI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Christina Darviri, Professor, National and Kapodistrian University of Athens
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: 472 /07-12-2023
Record Dates: First submitted 2024-11-11; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Psoriasis
Keywords: Psoriasis; Pythagorean self-awareness intervention; Stress management; Perceived stress; Sleep quality; Cognitive function; Hair Cortisol; Clinical samples
MeSH Terms: conditions — Psoriasis; Sleep Initiation and Maintenance Disorders | interventions — Health Promotion

STUDY DESIGN:
Intervention Model Description: A one-group pretest-posttest design, incorporating two pretest measurements (i.e., a double pretest) to enhance the methodological rigor. Specifically, participants were assessed twice prior to the intervention (using both questionnaires and devices) and once after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pretest T0 (No Intervention): Usual care
- Pretest T1 (No Intervention): Usual care
- Post-test T2 (Experimental): PSAI
  Interventions: Behavioral: Pythagorean Self-Awareness Intervention for stress management and health promotion

INTERVENTIONS:
Behavioral: Pythagorean Self-Awareness Intervention for stress management and health promotion — Pythagorean Self-Awareness is a holistic stress magement program that combines cognitive reconstruction and the implementation of the 6 pillars of life-style medicine depending on the targeted population.
  Other Names: PSAI
  Arms: Post-test T2

SUMMARY:
This one-arm, pilot, non-randomized, study was conducted at the Specialized Psoriasis Unit of Andreas Syggros Hospital in Athens, Greece. All participants were informed about the objectives and procedures of the study, and written informed consent was provided prior to participation. The study protocol was approved by the hospital's Scientific and Ethics Committee (protocol number: 472 /07-12-2023)and was in accordance with the Declaration of Helsinki.

DETAILED DESCRIPTION:
Pythagorean Self-Awareness Intervention (PSAI) to a sample of psoriasis patients. Primary aim was the reduction of perceived stress levels. Secondary aims were the enhancement of stress response (HRV), increase cortisol levels, improvement of sleep quality, adoption of healthy behaviors, emotional regulation (e.g., shame and anger), cognitive performance enhancement (e.g., visual-spatial memory, verbal learning, information processing speed), as well as improvements in body composition indices (e.g., weight, body mass index (BMI), intermuscular adipose tissue (IMAT), fat mass, and free fat mass).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of psoriasis
* Speaking and writing in Greek language

Exclusion Criteria:

* Use of oral corticosteroids
* Diagnosis of any serious mental disorder
* Drug addictions

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-12-04 (Actual); Primary Completion 2024-07-08 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS-14) | Two times before the intervention (with 1 month distance) and 4 months after baseline measurements
  To assess perceived stress, the Greek version of the PSS questionnaire was administered, which consists of 14 items, each graded on a 5-point Likert scale. More specifically, there are seven positive and seven negative items and the total score ranges from 0 to 56. Higher PSS scores indicate higher levels of perceived in the past month.
Hair cortisol | Two times before the intervention (with 1 month distance) and 4 months after baseline measurement
  Hair samples were collected from each participant twice prior to the intervention and once following the intervention. The samples were taken from the posterior vertex of the scalp. Cortisol levels were analyzed retrospectively by examining the hair segments. The proximal 1 cm segment closest to the scalp reflects cortisol secretion over the past month, while the second most proximal 1 cm segment represents cortisol production from the preceding month, and so on.

SECONDARY OUTCOMES:
Heart Rate Variability | Two times before the intervention (with 1 month distance) and 4 months after baseline measurement
  To collect HRV data via ECG, we utilized the NeXus hardware in combination with the BioTrace+ software (NeXus-10 version 2023; BioTrace+, Mind Media, Herten, the Netherlands). The NeXus system integrates HRV-BF with psychophysiological research and offers ECG data in both time and frequency domains using self-adhesive electrodes. The researcher manually initiated NeXus measurements at the start of the PPG data collection to ensure simultaneous acquisition of both PPG and ECG data.
Pittsburgh Sleep Quality Index | Two times before the intervention (with 1 month distance) and 4 months after baseline measurement
  Sleep quality was assessed using the Greek version of the PSQI questionnaire. The PSQI consists of 19 self-report questions, grouped into 7 components (subjective sense of sleep quality, awakening time, latent period, duration, usual sleep productivity, use of sleep medication and daytime dysfunction). The score ranges from 0 to 3, resulting in a total score ranging from 0=high sleep quality to 21=low sleep quality. A total score of > or = 5 indicates poor sleep
Healthy Life-style and Personal Control Questionnaire | Two times before the intervention (with 1 month distance) and 4 months after baseline measurement
  The healthy lifestyle and self-monitoring questionnaire consists of 26 items, which are divided into a 4-point Likert scale ranging from 1=never/rarely to 4= always. A higher score indicates increased health empowerment. Specifically, the HLPCQ is designed to assess one's degree of control over daily activities such as diet, daily schedule, physical activity, socialization and pessimistic thoughts
Cognitive assessment | Two times before the intervention (with 1 month distance) and 4 months after baseline measurement
  The standardized battery Brief Intentory for Cognitive Assessment(BICA) was used to assess cognitive functions in the participants. This memory assessment tool took about 15 minutes to complete is completed and included three categories of cognitive tests: The Normal Symbol Digital Modalities Test (SDMT), which measured information processing speed, the California Verbal Learning Test-II (CVLT-II), which assessed verbal memory and subsequent immediate recall. Finally, the third test concerned short visuospatial memory Test Revised (BVMTR), which assessed visual memory and immediate recall. Low scores indicated cognitive dysfunctions and cognitive decline. The specific tool for memory assessment has been proposed to help practitioners identify a potential cognitive dysfunction in humans.
Anger evaluation | Two times before the intervention (with 1 month distance) and 4 months after baseline measurement
  The STAXI questionnaire examines how individuals respond or behave when they feel angry. The Greek version of the 24-item STAXI was utilized. The items are rated on a four-point Likert-type scale (1 ¼ almost never to 4 ¼ almost always) three subscales: not expressing anger, expressing anger, controlling anger.
Shame, Guilt and Pride assessment | Two times before the intervention (with 1 month distance) and 4 months after baseline measurement
  The State Shame and Guilt Scale is a 15-item self-report questionnaire designed to assess shame, guilt and pride in response to a specific situation. Participants rate their responses on a 5-point Likert scale, ranging from "I don't feel that way at all" to "I feel very strongly that way".
Health Locus of Control (HLC) | Two times before the intervention (with 1 month distance) and 4 months after baseline measurement
  The HLC scale was employed to assess participants' beliefs regarding their perceived control over their health. This 18-item scale is divided into three subscales: HLC internal, HLC external, and HLC chance (denoted as HLC-1, HLC-2, and HLC-3, respectively). The internal HLC subscale measures the extent to which an individual believes they are responsible for their own health and well-being. The HLC external subscale assesses the degree to which individuals attribute their health to external factors, such as other people or societal influences. The HLC subscale reflects beliefs that health outcomes are governed by chance or random factors beyond the individual's control. Higher scores on each subscale indicate a stronger belief in the corresponding type of control (internal, external, or chance) as a determinant of health.

CONTACTS AND LOCATIONS:
Overall Officials: Christina Darviri, Professor, Study Director — Postgraduate Course of Stress Science & Health Promotion, NKUA, Greece
Locations (1):
- Andreas Syggros Hospital, Athens, Greece

IPD SHARING:
Plan to Share IPD: No
Upon request after publication

REFERENCES:
- [Background] Panagopoulou Z, Artemiadis AK, Chrousos GP, Darviri C, Anagnostouli MC. Pythagorean Self-Awareness Intervention for Multiple Sclerosis Patients: A Quasi-Experimental Pragmatic Trial. Arch Clin Neuropsychol. 2022 Jan 17;37(1):125-132. doi: 10.1093/arclin/acab044. PMID 34128954
- [Background] Psarraki EE, Bacopoulou F, Panagoulias E, Michou M, Pelekasis P, Artemiadis A, Chrousos GP, Darviri C. The effects of Pythagorean Self-Awareness Intervention on patients with major depressive disorder: A pilot randomized controlled trial. J Psychiatr Res. 2021 Jun;138:326-334. doi: 10.1016/j.jpsychires.2021.03.067. Epub 2021 Apr 13. PMID 33894540
- [Background] Gorgili K, Artemiadis A, Bacopoulou F, Karatzas P, Tigani X, Vlachakis D, Kokka I, Varvogli L, Chrousos GP, Darviri C. The Effects of Pythagorean Self-Awareness Intervention on Irritable Bowel Syndrome Patients: A Non-randomized Controlled Trial. Adv Exp Med Biol. 2021;1337:345-354. doi: 10.1007/978-3-030-78771-4_39. PMID 34972923
- [Background] Charalampopoulou M, Bacopoulou F, Syrigos KN, Filopoulos E, Chrousos GP, Darviri C. The effects of Pythagorean Self-Awareness Intervention on breast cancer patients undergoing adjuvant therapy: A pilot randomized controlled trial. Breast. 2020 Feb;49:210-218. doi: 10.1016/j.breast.2019.12.012. Epub 2019 Dec 20. PMID 31901782
- [Background] Athanasopoulou S, Simos D, Charalampopoulou M, Tentolouris N, Kokkinos A, Bacopoulou F, Aggelopoulou E, Zigkiri E, Chrousos GP, Darviri C, Gonos ES. Significant improvement of stress and aging biomarkers using a novel stress management program with the cognitive restructuring method "Pythagorean Self-Awareness Intervention" in patients with type 2 diabetes mellitus and healthy adults. Mech Ageing Dev. 2021 Sep;198:111538. doi: 10.1016/j.mad.2021.111538. Epub 2021 Jul 1. PMID 34217756